CLINICAL TRIAL: NCT02362477
Title: Telemental Health and Cognitive Processing Therapy for Female Veterans With Military-related PTSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Pacific Islands Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-10-1-1037; PT090552 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2015-02-04; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control CPT (Active Comparator): 'Cognitive Processing Therapy in-person. Cognitive Processing Therapy is delivered to female veterans and civilians, who have been diagnosed with PTSD, in-person.
  Interventions: Behavioral: Cognitive Processing Therapy in-person
- Experimental CPT via VTC (Experimental): 'Cognitive Processing Therapy through videoteleconference. Cognitive Processing Therapy is delivered to female veterans and civilians, who have been diagnosed with PTSD, through videoteleconference.
  Interventions: Behavioral: Cognitive Processing Therapy through videoteleconference

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy in-person — Cognitive Processing Therapy is delivered to female veterans and civilians, who have been diagnosed with PTSD, in-person.
  Other Names: CPT-NP
  Arms: Control CPT
Behavioral: Cognitive Processing Therapy through videoteleconference — Cognitive Processing Therapy is delivered to female veterans and civilians, who have been diagnosed with PTSD, through videoteleconference.
  Other Names: CPT-VTC
  Arms: Experimental CPT via VTC

SUMMARY:
The immediate objective of this project is to evaluate the clinical effectiveness of a telemental health modality (video-teleconferencing) for providing an evidence-based group intervention to female rural veterans, Reservists, National Guardsmen, and civilians suffering with PTSD. This study is an expansion, seeking to add a treatment arm of women, to an already CDMRP-funded study that completed in July 2014 treating male combat veterans with military-related PTSD. The long-term objective of this project is to disseminate an empirically sound TMH PTSD protocol for male and female veterans, Reserve and Guard that will extend the use of CPT to remote rural sites. It is hypothesized that using VTC, will be as effective as the in-person mode of service delivery for providing CPT.

DETAILED DESCRIPTION:
This expansion is a 4-year RCT, plus a 1 year no-cost extension, which provides a direct comparison of the VTC and in-person modalities using rigorous methodology and a sophisticated analysis of treatment equivalency in clinical and process outcome domains. Outcome domains include clinical and process outcomes. Approximately 154 female veterans, Reservists, National Guardsmen, or civilians with PTSD have been recruited from multiple VA clinical sites and community health centers (for N=110 completers). Consistent with the male combat veterans CPT study, prospective participants received a comprehensive assessment battery at baseline to determine eligibility. The exclusion criteria selected are consistent with large PTSD randomized clinical trials as well as research using the CPT protocol with military populations with PTSD. The treatment is delivered up to twice a week for up to 12 weeks by a doctoral level psychologist. Quality control procedures have been incorporated into the study's design to ensure integrity, fidelity and standard administration of the CPT intervention across both conditions. It is expected that the results from this project can be applied to other VA and military locations, where similar specialized PTSD clinical services are needed but unavailable due to geographic barriers.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of current PTSD established by the Clinician-Administered PTSD Scale (CAPS) and
* a stable psychotropic medication regimen for a minimum of 45 days prior to study entry for those taking such medications.

Exclusion Criteria:

* significant cognitive impairment or history of organic mental disorder,
* active psychotic symptoms/disorder,
* active homicidal or suicidal ideation,
* current substance dependence, and
* unwillingness to refrain from substance abuse during treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS-IV) | 6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A. Morland, Psy.D., Principal Investigator — VA Pacific Islands Healthcare System
Locations (1):
- VA Pacific Islands Healthcare System, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Glassman LH, Mackintosh MA, Wells SY, Wickramasinghe I, Walter KH, Morland LA. Predictors of Quality of Life Following Cognitive Processing Therapy Among Women and Men With Post-Traumatic Stress Disorder. Mil Med. 2020 Jun 8;185(5-6):e579-e585. doi: 10.1093/milmed/usz474. PMID 32077948